CLINICAL TRIAL: NCT03826992
Title: A Phase I Study of Venetoclax Combined With Vyxeos (CPX-351) for Children, Adolescents and Young Adults With Relapsed or Refractory Acute Leukemia
Brief Title: Venetoclax Combined With Vyxeos (CPX-351) for Participants With Relapsed or Refractory Acute Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V2-MA-1801
Record Dates: First submitted 2019-01-09; First posted 2019-02-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Leukemia
Keywords: relapsed; refractory; Vyxeos; Venetoclax; acute myeloid leukemia; acute myeloid leukemia, childhood; mixed-lineage leukemia (MLL); AML; CPX-351; Venclexta; Histone-lysine N-methyltransferase 2A (KmT2A)
MeSH Terms: conditions — Leukemia; Recurrence; Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; CPX-351; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax and Vyxeos combination (Experimental): Venetoclax will be given orally on Days per the assigned dose level. A single course consisting of 3 doses of Vyxeos and 7-21 doses of venetoclax depending on the assigned dose level will be administered to participants in this study. Vyxeos will be administered by central venous catheter over 90 minutes on Day 1, 3, and 5.
  Venetoclax is given daily by mouth per assigned dose level.
  Interventions: Drug: Vyxeos; Drug: Venetoclax

INTERVENTIONS:
Drug: Vyxeos — Vyxeos Dose: daunorubicin 44 mg/m2 and cytarabine 100 mg/m2 administered via intravenous infusion over 90 minutes on Days 1, 3, and 5.
  Other Names: cytarabine and daunorubicin liposome, CPX-351
Drug: Venetoclax — Venetoclax Dose:
  1. Dose Level 0 - weight based daily dosing for 21 days
  2. Dose Level -1 - weight based daily dosing for 14 days
  3. Dose Level -2- weight based daily dosing for 10 days
  4. Dose Level -3- weight based daily dosing for 7 days
  Other Names: Venclexta

SUMMARY:
This study evaluates the safety and tolerability of combining venetoclax with Vyxeos (CPX-351) in pediatric and young adult patients with acute leukemia that has come back or not responded to treatment.

DETAILED DESCRIPTION:
This is a single-institution Phase I pilot study designed to test the safety and tolerability of combining venetoclax with Vyxeos (CPX-351, cytarabine and daunorubicin liposome) for the treatment of relapsed/refractory acute leukemia in young patients. Subjects will receive a single course of study therapy consisting of daily, oral or crushed venetoclax at an assigned dose level with a 3-day ramp-up to target dose and Vyxeos administered intravenously at the established dose on Days 1, 3, and 5. In addition to safety and tolerability, the overall response rate to these therapies will be estimated. Pharmacokinetic (PK) analysis will also be conducted to define the drug clearance of venetoclax in this combination.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 Year to 39 Years
* Diagnosis of one of the following:

  * Acute myeloid leukemia (AML), any subtype except

    * Patients with acute promyelocytic leukemia (APML) are NOT eligible
    * Patients with ML-DS are NOT eligible
  * Myeloid sarcoma
  * Acute leukemia of ambiguous lineage (ALAL)

    * Acute undifferentiated leukemia (AUL)
    * T/myeloid mixed phenotype acute leukemia (MPAL)
    * B/myeloid MPAL
    * MPAL with KMT2A-rearrangement MPAL with t (9;22) are NOT eligible
  * T-cell acute lymphoblastic leukemia (T ALL)
  * Early thymocyte precursor (ETP) ALL
  * KMT2A-rearranged ALL
* Disease Status

  * Relapsed/Refractory AML, MPA, and AUL
  * Untreated therapy related AML
  * Relapsed/Refractory KMT2A-rearranged ALL, T-cell ALL, ETEP ALL
* Karnofsky/Lanksy performance level score of greater than or equal to 50 percent.
* Prior therapy requirements

  * Fully recovered from acute toxicities of Hematopoietic Stem Cell Transplant (HSCT) or Anthracycline Exposure
  * 14 days must have elapsed since the completion of systemic cytotoxic therapy other than hydroxyurea, decitabine or azacitidine
  * 2 weeks must have elapsed for local palliative radiotherapy (RT); 6 months must have elapsed if prior craniospinal RT or if 50% radiation of pelvis, and at least 6 weeks must have elapsed if other substantial bone marrow radiation
* Adequate renal, liver, cardiac, and central nervous system (CNS) function

Exclusion Criteria:

* Diagnosis of one of the following:

  * Myeloid Leukemia associated with Down Syndrome (ML-DS)
  * Acute Promyelocytic Leukemia (APML)
  * Acute leukemia with CNS status 3 involvement
  * Philadelphia chromosome t(9;22) positive leukemia (Ph+ ALL, AML, MPAL, or AUL)
  * Fanconi Anemia, Shwachman-Diamond syndrome, or any other bone marrow failure syndrome or DNA repair disorder
  * Wilson's Disease or other copper-metabolism disorder
* Pregnant or breastfeeding
* Uncontrolled infection
* Received greater than 13.6 Gray (Gy) prior radiation to the mediastinum
* Receipt of growth factors within 7 days prior to enrollment
* Currently receiving another investigational drug
* Currently receiving anti-cancer agents (with the exception of intrathecal (IT) agents or hydroxyurea)
* Unable to comply with the safety monitoring requirements of the study

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of combining venetoclax and Vyxeos (dose limiting toxicities) | 28 days
  If 2 or more participants have dose limiting toxicities at a given dose level, the maximum tolerated dose will have been exceeded.
Treatment related toxicities | 60 days
  Number of related adverse events

SECONDARY OUTCOMES:
Disease response | 42 days
  Estimate of overall response rate (ORR) defined as (CR/CRi/CRp).
Cancer therapeutics-related cardiac dysfunction (CTRCD) in patients who have previously received anthracyclines | 60 days
  Measured by echocardiogram (ECHO)

CONTACTS AND LOCATIONS:
Overall Officials: John Perentesis, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cincinnati Children's Cancer and Blood Diseases Institute — http://www.cincinnatichildrens.org/research/divisions/c/cbdi/default/
- See also: Cincinnati Children's Hospital Oncology Division — http://www.cincinnatichildrens.org/research/divisions/o/oncology/default/
- See also: Leukemia and Lymphoma Program — http://www.cincinnatichildrens.org/service/l/leukemia-lymphoma/clinical-trials/